CLINICAL TRIAL: NCT03492424
Title: Ablative Therapy in the Management of Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 1702017952 prev. 1702018011
Record Dates: First submitted 2018-03-30; First posted 2018-04-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; cryotherapy; focal therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Focal therapy for prostate cancer: All men >18 years of age undergoing focal therapy for primary or salvage treatment of prostate cancer will be included. Men who had received prior focal therapy are also eligible for inclusion.
  The purpose of this study is collect observational data regarding patterns of care and outcomes of focal therapies for prostate cancer, including but not limited to: high-intensity focused ultrasound (HIFU), cryotherapy, focal laser ablation, irreversible electroporation, photodynamic therapy, and brachytherapy.
  Interventions: Device: cryotherapy

INTERVENTIONS:
Device: cryotherapy — Subjects will receive focal cryotherapy for treatment of prostate cancer

SUMMARY:
The purpose of this study is collect observational data regarding patterns of care and outcomes of focal therapies for prostate cancer, including but not limited to: high-intensity focused ultrasound (HIFU), cryotherapy, focal laser ablation, irreversible electroporation, photodynamic therapy, and brachytherapy.

DETAILED DESCRIPTION:
Through the use of a pro- and retrospective registry, the investigators will collect information on patient characteristics including age, co-morbidities, imaging and biopsy information, and prior treatments. Information on treatment details will also be captured, including treatment time, anesthesia delivered, and length of stay, when applicable. Oncologic outcomes including PSA, post-treatment biopsy and imaging data, need for re-treatment, and survival outcomes will also be captured. Safety outcomes will be captured using the Clavien-Dindo classification scale, and additional specific GU complications will be recorded, which include urinary retention, urethral stricture, recto-urethral fistula, osteomyelitis, and urinary tract infection. Finally, the investigators will capture functional outcomes using health related quality of life questionnaires including the EPIC questionnaire, IIEF-5, MSHQ-EjD, and IPSS.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Undergoing focal therapy for primary or salvage treatment of prostate cancer, or
* Have received prior focal therapy

Exclusion Criteria:

* Clinically-evident metastatic disease
* Unable to fill out an English-language questionnaire

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are generally healthy men diagnosed with prostate cancer, undergoing focal therapy for treatment of prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2032-03-02 (Estimated); Study Completion 2039-09-02 (Estimated)

PRIMARY OUTCOMES:
Prostate biopsy Gleason grade | 12 months
  Will be obtained through patient biopsy pathology results

SECONDARY OUTCOMES:
Patient characteristics/demographics | 12 months
  Will be obtained through patient medical history in electronic health record
MRI PI-RAD grade | 12 months
  Will be obtained through patient MRI radiology results
Lab results - PSA level | 12 months
  Will obtain patient PSA (ng/mL) through laboratory (blood) results
Patient-reported quality of life: EPIC-26 | 12 months
  Expanded Prostate Cancer Index Composite (short form) questionnaire to assess quality of life
Patient-reported quality of life: IIEF-5 | 12 months
  The International Index of Erectile Function questionnaire to assess erectile function
Patient-reported quality of life: MSHQ-EjD | 12 months
  Male Sexual Health questionnaire to assess ejaculatory function
Patient-reported quality of life: IPSS | 12 months
  International Prostate Symptom Score questionnaire to assess urinary function and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Tim McClure, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No